CLINICAL TRIAL: NCT01967459
Title: Effects of High and Low Dose Vitamin D Suppletion on Postprandial Leukocyte Activation, Oxidative Stress and Vascular Function in Healthy Overweight and Obese Females
Brief Title: Effects Vitamin D Suppletion on Postprandial Leukocyte Activation
Acronym: DOSFEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, M.A. de Vries, MD, Sint Franciscus Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL44804.101.13
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Atherosclerosis; Oxidative Stress; Leukocyte Activation Disorder
MeSH Terms: conditions — Atherosclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose vitamin D (Active Comparator): Volunteers assigned to this arm will receive a single dose of oral cholecalciferol 300 000 IU, in the form of 3 ml D-cura drink 100 000 IU/ml
  Interventions: Drug: Cholecalciferol
- Low dose vitamin D (Active Comparator): Volunteers assigned to this arm will receive a single dose of oral cholecalciferol 75000 IU, in the form of 3 ml D-cura drink 25 000 IU/ml
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Single dose D-cura cholecalciferol drink 100 000 IU/ml, in total 300 000 IU (=3ml)
  Other Names: D-cura
  Arms: High dose vitamin D
Drug: Cholecalciferol — Single dose D-cura cholecalciferol drink 250 000 IU/ml, in total 75 000 IU (=3ml)
  Other Names: D-cura
  Arms: Low dose vitamin D

SUMMARY:
Administration of vitamin D will have a beneficial effect on postprandial leukocyte activation, oxidative stress and arterial stiffness in vitamin D deficient females. High doses of vitamin D may have a more pronounced effect than low doses.

DETAILED DESCRIPTION:
Rationale: Postprandial lipemia, known to be associated with acute leukocyte activation, impairs endothelial function and promotes atherosclerosis. Deficiency of vitamin D is associated with increased cardiovascular risk, but the precise mechanism is still unclear. A recent pilot study performed in our laboratory showed improved postprandial vascular function by pulse wave analysis and decreased postprandial leukocyte activation after vitamin D supplementation. Interestingly, the effects on leukocyte activation were solely found in females.

Hypothesis: The beneficial effects of vitamin D administration on postprandial leukocyte activation are mediated by suppression of oxidative stress. High doses of vitamin D may have a more pronounced effect than low doses.

Objective: To estimate the effect sizes of different doses of vitamin D on postprandial leukocyte activation markers, oxidative stress and arterial stiffness in vitamin D deficient females.

Study design: Randomized, double blind pilot study. Study population: Premenopausal overweight and obese female volunteers with proven vitamin D deficiency, ≥ 18 years of age.

Intervention: Two oral fat load tests (OFLTs) will be performed. After the first OFLT, volunteers will be randomly assigned to receive a single low dose (75 000 IU) or high dose (300 000 IU) of cholecalciferol drink. One week later the OFLT will be repeated.

Main study parameters/endpoints: Postprandial leukocyte activation, oxidative stress parameters and arterial augmentation index.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The use of a single dose of 300 000 IU of cholecalciferol has been established to be a safe and effective way to correct vitamin D deficiency. Volunteers will be hospitalized on 2 different days (day 1, day 8) for approximately nine hours each day and receive an oral fat load. Cholecalciferol will be administered once. Volunteers will be instructed not to take vitamin D supplements during the study up until 3 months after the study. The volunteers' general practitioner will be informed on their participation. A total of 222ml (111ml for each postprandial test) of blood will be drawn. Volunteers will be allowed to drink only water during the tests. There is a theoretical risk of hypercalcemia but no excessive risk is involved. Volunteers receive 250 euros for full participation. Furthermore, volunteers will be told and given advice if they turn out to suffer from hyperlipidemia or any other condition.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older;
* Pre-menopausal;
* BMI ≥25.0 kg/m2;
* Vitamin D deficiency, defined by a 25-hydroxyvitamin D level of <30ng/ml;
* Use of oral contraceptives.

Exclusion Criteria:

* The use of any kind of medication except oral contraceptives;
* Smoking;
* Pregnancy;
* Participation in a clinical study less than 6 months before inclusion;
* The use of (multi)vitamin supplements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
effect of vitamin D on leukocyte cluster of differentiation antigen 11b expression | 2, 4, 6 and 8 hours postprandial
  the differential effect of 75 000 IU low dose vs. 300 000 IU high dose vitamin D on postprandial leukocyte activation markers cluster of differentiation antigen 11b

SECONDARY OUTCOMES:
Effect of vitamin D on oxidative stress | 2,4,6 and 8 hours postprandial
  the differential effect of 75 000 IU low dose vs. 300 000 IU high dose vitamin D on oxidative stress
Effect of vitamin D on vascular function | 0,2,6,8 and 8 hours postprandial
  the differential effect of 75 000 IU low dose vs. 300 000 IU high dose vitamin D on vascular function (Pulse Wave Velocity and Augmentation Index)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castro Cabezas, MD, PhD, Study Chair — Sint Franciscus Gasthuis
Locations (1):
- Sint Franciscus Gasthuis, Rotterdam, South Holland, Netherlands